CLINICAL TRIAL: NCT01795573
Title: Phase I Trial of Ex-vivo Expanded Donor Regulatory T Cells for Prevention of Acute Graft-Versus-Host Disease
Brief Title: Ex-vivo Expanded Donor Regulatory T Cells for Prevention of Acute Graft-Versus-Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-17263
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Graft Versus Host Disease
Keywords: GVHD; AML; ALL; MDS; CLL; NHL; HL; MM
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cultured Treg cells (Other): Co-culturing of recipient dendritic cells and donor Treg cells given prior to allogeneic stem cell transplant
  Interventions: Biological: Cultured Treg cells

INTERVENTIONS:
Biological: Cultured Treg cells — Co-culturing of recipient dendritic cells and donor Treg. Treg administration will occur 2 days before the allogeneic stem cell transplant (i.e. day -2 with reference of day 0 as stem cell infusion date).

SUMMARY:
Clinical trial of allospecific regulatory t cells (Tregs) for prevention of acute graft-versus-host disease (GVHD) in human leukocyte antigen (HLA) identical sibling transplants.

DETAILED DESCRIPTION:
To evaluate the safety of sirolimus based immune suppression and ex-vivo expanded donor regulatory T cells for the prevention of acute graft-versus-host disease following allogeneic hematopoietic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnoses:

  a. Hematologic malignancies - Acute myelogenous leukemia (AML), acute lymphoblastic leukemia (ALL), myelodysplastic syndrome (MDS), chronic lymphocytic leukemia (CLL), non-Hodgkin lymphoma (NHL), Hodgkin lymphoma (HL), multiple myeloma (MM) - in complete remission (CR). Complete remission is defined per morphologic, cytogenetic, FISH, molecular, and radiographic imaging studies appropriate for each condition listed.
  * AML, ALL: Normal values for absolute neutrophil count (>1000/microL) and platelet count (>100,000/microL); Absence of extramedullary leukemia; Less than 5 percent blast cells present in the bone marrow
  * MDS: Bone marrow with ≤5 percent myeloblasts with normal maturation of all cell lines; Peripheral blood demonstrates hemoglobin ≥11 g/dL, platelets ≥100 x 10^9/L, neutrophils ≥1 x 10^9/L, and no circulating blasts
  * CLL: Absence of constitutional symptoms attributable to CLL; No lymph nodes >1.5 cm in diameter on computed tomography; No hepatomegaly or splenomegaly by computed tomography; Absolute neutrophil count >1500/microL; Platelet count >100,000/microL; No clonal lymphocytes in the peripheral blood by immunophenotyping; Bone marrow with no evidence of clonal CLL (by flow cytometry and/or immunohistochemistry
  * NHL: No clinical evidence of disease or disease-related symptoms; Typically FDG-avid lymphomas: a post-treatment residual mass of any size is permitted as long as it is PET negative; Variably FDG-avid lymphoma/FDG avidity unknown: all lymph nodes normal size by CT; Spleen and liver non-palpable and without nodules; If pretreatment bone marrow biopsy was positive, repeat bone marrow biopsy must be negative; if morphologically indeterminate, immunohistochemistry should be negative If pretreatment bone marrow biopsy was positive, repeat bone marrow biopsy must be negative; if morphologically indeterminate, immunohistochemistry should be negative
  * HL: No clinical evidence of disease or disease-related symptoms; A post-treatment residual mass of any size is permitted as long as it is PET negative; Spleen and liver must be non-palpable and without nodules; If a pre-treatment bone marrow biopsy was positive, an adequate bone marrow biopsy from the same site must be cleared of infiltrate; if this is indeterminate by morphology, immunohistochemistry should be negative
  * MM: Absence of monoclonal protein in serum and urine by immunofixation with no current evidence of soft tissue plasmacytoma; Bone marrow aspirate and biopsy must demonstrate less than 5 percent clonal plasma cells; In patients who lack measurable M proteins in the serum and urine being monitored using the FLC levels, the definition of CR requires a normalization of the free light chain (FLC) ratio in addition to the above criteria
  * MDS: May have achieved CR through either hypomethylating agent therapy, induction chemotherapy, or other therapy
  * MDS: Low/intermediate-1 IPSS risk category patients are eligible only if they have failed prior therapy or are transfusion-dependent
* Peripheral blood white blood count (WBC) greater than 2,000 per microliter (required for collection of dendritic cell precursors)
* Adequate vital organ function: Left ventricular ejection fraction (LVEF) ≥ 45% by multigated acquisition (MUGA) scan or echocardiogram; Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and diffusing lung capacity oxygenation (DLCO) ≥ 50% of predicted values on pulmonary function tests; Transaminases (AST, ALT) < 3 times upper limit of normal values; Creatinine clearance ≥ 50cc/min
* Infectious disease criteria:

  * No active infection; infection controlled with antimicrobial therapy is not excluded
  * HIV negative by ELISA or reverse transcription polymerase chain reaction (RT-PCR) [if ELISA is positive and RT-PCR is negative, the ELISA is considered false positive]
  * Hepatitis B and C negative by serology or RT-PCR
  * Must complete full screening panel: HIV 1, 2 serology and RT-PCR; human T cell lymphotropic virus types 1/2 (HTLV-1/2) serology; rapid plasma reagin (RPR) serology; Epstein-Barr virus (EBV) serology; Cytomegalovirus (CMV) serology; herpes simplex virus (HSV) serology; Varicella-. Zoster Virus (VZV) serology
* Performance status: Karnofsky Performance Status Score ≥ 60%.
* Agreement to utilize effective contraceptive methods during the study (for one year)
* Eligible donors will include siblings age ≥ 18 matched with the recipient at HLA-A, B, C, and DRB1

Exclusion Criteria:

* Antithymocyte globulin (ATG) as part of the conditioning regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-10-29 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Maximally Tolerated dose (MTD) | Up to 1 year
  MTD of donor Treg in combination with standard dose SIR/TAC immune suppression. The occurrence of dose-limiting toxicity in >= 33% serves as the boundary for the MTD of donor Treg.

SECONDARY OUTCOMES:
Acute GVHD incidence | Up to day 100
  Clinical evidence of acute GVHD will be recorded per standard grading scheme. GVHD grade will be reported weekly from day 0-100 both for site-specific involvement, as well as an overall composite score.
Relapse Free Survival | Up to 1 year
  Defined as time from transplantation (day 0 as day of stem cell infusion per standard nomenclature) to relapse or death from any cause.
Non-relapse Mortality | Up to 1 year
  Defined as mortality while underlying malignancy is in remission.
Overall Survival (OS) | Up to 1 year
  Defined as time from transplantation (day 0 as day of stem cell infusion per standard nomenclature) to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pidala, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- H Lee Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: H. Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org/